CLINICAL TRIAL: NCT02105727
Title: A Before After Comparison of the Effectiveness of a Community-based Salt Reduction Program Done in Lithgow, Australia
Brief Title: Changing Population Salt Consumption in Lithgow, Australia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: New South Wales Health (Unknown); New South Wales Food Authority (Unknown); Australian Food and Grocery Council (Unknown); National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Professor Bruce Neal, Professor, The George Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014079
Record Dates: First submitted 2014-03-30; First posted 2014-04-07 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Blood Pressure; Hypertension; Cardiovascular Disease
Keywords: Dietary sodium; Urinary sodium excretion; Urinary iodine excretion
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Salt reduction (Experimental): Community-based salt reduction
  Interventions: Behavioral: Community-based salt reduction

INTERVENTIONS:
Behavioral: Community-based salt reduction
  Other Names: Salt-substitute; Education; Smartphone application - FoodSwitch/Saltswitch

SUMMARY:
The objective of this study is to determine whether a community-based salt reduction program can reduce average salt consumption levels. Baseline levels of salt consumption were measured in 2011, the salt reduction program was then implemented, and now in 2014 investigators are remeasuring salt consumption levels in the community. The hypothesis investigators are testing is that the salt reduction program will have led to a change in salt consumption levels between 2011 and 2014. The study is being done in Lithgow, a regional town in New South Wales , Australia.

DETAILED DESCRIPTION:
The primary objective of this project is to determine whether there have been changes in average salt consumption levels in the Lithgow population from 2011 to 2014. The primary null hypothesis to be tested is that there will be no difference between the mean 24-hour urinary sodium excretion levels between 2011 and 2014.

The sample of 419 individuals with 24-hour urine samples in the baseline survey and 600 individuals in the follow-up survey will provide 80% power to detect a difference of 0.7 g/day salt between the mean levels of excretion before and after the intervention. There will be more than 95% power to detect a difference of 1.0 g/day salt or greater.

ELIGIBILITY:
Inclusion Criteria:

* All adults over the age of 20 years residing in the Lithgow area are eligible
* No exclusion based on inter-current illness, use of medications or any other aspect of demography or personal history.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 991 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion (mmol/l) | up to 4 years
  A single 24-hour urine collection will be obtained with the first voided urine upon waking on the day of collection being discarded and participants then collecting all voided urine up to and including the first void the following morning. The times at the beginning and the end of urine collection are recorded.

SECONDARY OUTCOMES:
Sources of sodium | up to 4 years
  The multiple pass 24-hour dietary recall is used to determine all food and beverages consumed from midnight to midnight on the day before the interview, this method has been described in detail by prior reports. Food model booklets are used to assist with the reporting of quantity and prompts provided by interviewers are used to probe for complete food descriptions, variable recipe ingredients, and food preparation including salt added during cooking and at the table. Dietary data are entered into the nutrient analysis package FoodWorks Professional version 7. The food coding guidelines are used to code each food and beverage into major, sub-major and minor food categories.
Knowledge, attitudes and behaviors towards salt intake | up to 4 years
  The measurement of knowledge attitude and behaviors towards salt is based upon a questionnaire adapted from the World Health Organization/Pan American Health Organization protocol for population level sodium determination. The questionnaire contains nine questions; four related to knowledge of personal consumption, recommended daily intake and possible harmful effects of salt and five assessing attitudes and behaviors to lowering salt intake.

OTHER OUTCOMES:
Urinary iodine excretion (ug/l) | up to 4 years
  UIE will be assessed in the spot urine samples of females aged 20-45 years old. The measurement will be completed by using ammonium persulfate digestion prior to Sandell-Koltoff reaction in a microtitre plate format.

CONTACTS AND LOCATIONS:
Locations (1):
- The George Institute for Global Health, Camperdown, New South Wales, Australia

REFERENCES:
- [Background] Land MA, Webster J, Christoforou A, Johnson C, Trevena H, Hodgins F, Chalmers J, Woodward M, Barzi F, Smith W, Flood V, Jeffery P, Nowson C, Neal B. The association of knowledge, attitudes and behaviours related to salt with 24-hour urinary sodium excretion. Int J Behav Nutr Phys Act. 2014 Apr 4;11(1):47. doi: 10.1186/1479-5868-11-47. PMID 24708561
- [Result] Land MA, Webster J, Christoforou A, Praveen D, Jeffery P, Chalmers J, Smith W, Woodward M, Barzi F, Nowson C, Flood V, Neal B. Salt intake assessed by 24 h urinary sodium excretion in a random and opportunistic sample in Australia. BMJ Open. 2014 Jan 16;4(1):e003720. doi: 10.1136/bmjopen-2013-003720. PMID 24440795
- [Result] Land MA, Jeffery P, Webster J, Crino M, Chalmers J, Woodward M, Nowson C, Smith W, Flood V, Neal B. Protocol for the implementation and evaluation of a community-based intervention seeking to reduce dietary salt intake in Lithgow, Australia. BMC Public Health. 2014 Apr 14;14:357. doi: 10.1186/1471-2458-14-357. PMID 24731226
- [Derived] Land MA, Wu JH, Selwyn A, Crino M, Woodward M, Chalmers J, Webster J, Nowson C, Jeffery P, Smith W, Flood V, Neal B. Effects of a community-based salt reduction program in a regional Australian population. BMC Public Health. 2016 May 11;16:388. doi: 10.1186/s12889-016-3064-3. PMID 27169380